CLINICAL TRIAL: NCT05277636
Title: Acute Effects of R- and S-MDMA in Healthy Subjects
Acronym: R-S-MDMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2021-02386
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: 5-period random order, placebo-controlled, double-blind cross-over study with four active substance conditions and placebo:
  1. MDMA (125 mg), 2. S-MDMA (125 mg), 3. R-MDMA (125 mg), 4. R-MDMA (250 mg), 5. Placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 125 mg MDMA (Experimental): MDMA (125 mg)
  Interventions: Drug: 3,4-methylenedioxymethamphetamine
- 125 mg S-MDMA (Experimental): S-MDMA (125 mg)
  Interventions: Drug: S-3,4-methylenedioxymethamphetamine
- 125 mg R-MDMA (Experimental): R-MDMA (125 mg)
  Interventions: Drug: R-3,4-methylenedioxymethamphetamine (125 mg)
- 250 mg R-MDMA (Experimental): R-MDMA (250 mg)
  Interventions: Drug: R-3,4-methylenedioxymethamphetamine (250 mg)
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 3,4-methylenedioxymethamphetamine — A dose of 125 mg racemic MDMA will be administered.
  Other Names: MDMA
  Arms: 125 mg MDMA
Drug: S-3,4-methylenedioxymethamphetamine — A dose of 125 mg enantiomeric S-MDMA will be administered.
  Other Names: S-MDMA
  Arms: 125 mg S-MDMA
Drug: R-3,4-methylenedioxymethamphetamine (125 mg) — A dose of 125 mg enantiomeric R-MDMA will be administered.
  Other Names: R-MDMA
  Arms: 125 mg R-MDMA
Drug: R-3,4-methylenedioxymethamphetamine (250 mg) — A dose of 250 mg enantiomeric R-MDMA will be administered.
  Other Names: R-MDMA
  Arms: 250 mg R-MDMA
Other: Placebo — Placebo (Mannitol)
  Arms: Placebo

SUMMARY:
Racemic ±3,4-methylenedioxymethamphetamine (MDMA) is a psychoactive substance and prototypical empathogen acutely inducing feelings of heightened mood, empathy, trust and closeness to others. These acute subjective effects of MDMA may be helpful to assist psychotherapy and MDMA is currently investigated in phase 3 trials as a possible treatment in post-traumatic stress disorder.

DETAILED DESCRIPTION:
MDMA is a racemic substance containing equal amounts of the enantiomers S(+)- and R(-)-MDMA. Preclinical research indicates that S-MDMA mainly releases dopamine, norepinephrine, serotonin, and oxytocin while R-MDMA may act more directly on 5-HT2A receptors and release prolactin. Animal studies also indicate that the two enantiomers act synergistically to produce the subjective effects of MDMA and that S-MDMA is mainly responsible for psychostimulation while R-MDMA may have fewer adverse effects and have greater prosocial effects. However, acute effects of S- and R-MDMA have never been validly examined in a human study. Therefore, the present study compares acute responses to R-MDMA, S-MDMA, MDMA, and placebo in a cross-over study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years.
2. Understanding of the German language.
3. Understanding the procedures and the risks that are associated with the study.
4. Participants must be willing to adhere to the protocol and sign the consent form.
5. Participants must be willing to refrain from taking illicit psychoactive substances during the study.
6. Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
7. Participants must be willing not to drive a traffic vehicle or to operate machines within 48 h after substance administration.
8. Willing to use double-barrier birth control throughout study participation.
9. Body mass index between 18-29 kg/m2.

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder in first-degree relatives, not including psychotic disorders secondary to an apparent medical reason, e.g. brain injury, dementia, or lesions of the brain.
4. Hypertension (SBP>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Illicit substance use (not including cannabis) more than 20 times or any time within the previous month
6. Pregnant or nursing women.
7. Participation in another clinical trial (currently or within the last 30 days).
8. Use of medications that may interfere with the effects of the study medications.
9. Tobacco smoking (>10 cigarettes/day).
10. Consumption of alcoholic drinks (>15 drinks/week).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-01-13 (Actual); Study Completion 2024-01-13 (Actual)

PRIMARY OUTCOMES:
Subjective effects I | 18 months
  5 Dimensions of Altered States of Consciousness (5D-ASC) consisting of 94 items to be rated on a visual analog scale (0-100 mm), with higher values indicating stronger effects with higher scores representing more intense effects. Assessed once on each study day
Subjective effects II | 18 months
  Stimulation on the Visual Analog Scales (VAS) assessing the intensity and duration of the stimulant effect on a scale from 0 - 100 percent with higher scores representing more intense effects. Assessed 18 times on each study day

SECONDARY OUTCOMES:
Autonomic effects I | 18 months
  Assessed 18 times on each study day via systolic and diastolic blood pressure
Autonomic effects II | 18 months
  Assessed 18 times on each study day via heart rate
Autonomic effects III | 18 months
  Assessed 18 times on each study day via tympanic body temperature
Adverse effects | 18 months
  Assessed 3 times on each study day with the list of complaints (LC)
Mood after study day I | 18 months
  Assessed once 3 days after administration via the Beck Depressionindex questionnaire (BDI) with low values indicating normal mood and high values indicating severe depression
Mood after study day II | 18 months
  Assessed once 3 days after administration via Symptom checklist 90R (SCL-90R) to evaluate a number of different psychological symptoms.
Mood after study day III | 18 months
  Assessed once 3 days after administration via list of complaints (LC)
Mood after study day IV | 18 months
  Assessed once 3 days after administration via adjective mood rating scale (AMRS)
Plasma levels of cortisol | 18 months
  Assessed 3 times on each study day
Plasma levels of prolactin | 18 months
  Assessed 3 times on each study day
Plasma levels of oxytocin | 18 months
  Assessed 4 times on each study day
Plasma levels of vasopressin | 18 months
  Assessed 4 times on each study day
Plasma levels of S-MDMA | 18 months
  Assessed 17 times on each study day
Plasma levels of R-MDMA | 18 months
  Assessed 17 times on each study day
Plasma levels of S-MDA | 18 months
  Assessed 17 times on each study day
Plasma levels of R-MDA | 18 months
  Assessed 17 times on each study day
Additional subjective effects I | 18 months
  Visual Analog Scales (VAS) assessing the intensity and duration of subjective effects on a scale from 0 - 100 percent with higher scores representing more intense effects. Assessed 18 times on each study day
Additional subjective effects II | 18 months
  Adjective Mood Rating Scale (AMRS) assesses the occurrence and intensity of 60 moods on a 4-point Likert scale ranging from "not at all" to "extremely" assessed 4 times on each study day
States of Consciousness Questionnaire | 18 months
  Assesses the emergence and intensity of phenomenons occurring in altered states of consciousness on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely") once on each study day
Spiritual Realms Questionnaire | 18 months
  Assesses the spiritual phenomenons elicited by psychedelic substances through 11 main questions to be answered on a total of 65 sub-ordered 100mm visual analog scales once on each study day
Psychological Insight Questionnaire | 18 months
  Assesses the degree of psychological insight caused by a psychedelic experience through 14-items to be answered on a 6-point Likert scale ranging from 0 ("not at all") to 5 ("extremely") once on each study day
NEO-Five-Factor-Inventory (NEO-FFI) | Baseline
  The NEO-FFI is a self-description questionnaire with 60 items for the measurement of the "big five": neuroticism, extraversion, openness, agreeableness, and consciousness. It uses a 5-point Likert scale ranging from "completely disagree" to "fully agree".
Freiburger Personality Inventory (FPI-R) | Baseline
  The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Saarbrücker Personality Questionnaire (SPF) | Baseline
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
HEXACO personality inventory | Baseline
  The HEXACO personality inventory is a six-dimensional model of human personality with 100 items.The six factors are: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness and Openness to Experience.
Defense Style Questionnaire (DSQ-40) | Baseline
  The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital Basel, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Straumann I, Avedisian I, Klaiber A, Varghese N, Eckert A, Rudin D, Luethi D, Liechti ME. Acute effects of R-MDMA, S-MDMA, and racemic MDMA in a randomized double-blind cross-over trial in healthy participants. Neuropsychopharmacology. 2024 Dec;50(2):362-371. doi: 10.1038/s41386-024-01972-6. Epub 2024 Aug 23. PMID 39179638